CLINICAL TRIAL: NCT07113483
Title: Randomized, Double-Blind, 2x2 Factorial Trial of Remimazolam vs. Midazolam on Sedation and Early Cognitive Outcomes in Patients Undergoing Traumatic or Non-Traumatic Orthopedic Surgery With Regional Anesthesia
Brief Title: Remimazolam vs. Midazolam for Sedation and Cognitive Outcomes in Orthopedic Surgery
Acronym: REMIND-ORTHO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Romanian Society for Enteral and Parenteral Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35782025
Record Dates: First submitted 2025-07-17; First posted 2025-08-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Cognitive Dysfunction; Orthopedic Procedures; Postoperative Pain Management; Hip Fracture
Keywords: Remimazolam; Midazolam; Regional Anesthesia; Sedation; Cognitive dysfunction; Elderly patients; Trauma
MeSH Terms: conditions — Postoperative Cognitive Complications; Hip Fractures; Cognitive Dysfunction; Wounds and Injuries | interventions — Midazolam; Injections, Intravenous; Powders; remimazolam

STUDY DESIGN:
Intervention Model Description: Study medications (Remimazolam and Midazolam) will be prepared in identical syringes by a pharmacist not involved in patient care or outcome assessment. Both participants and clinical staff (anesthesiologists, nurses, outcome assessors) will be blinded to treatment allocation. Emergency unblinding is allowed only in the event of severe adverse events.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study medications (Remimazolam and Midazolam) will be prepared in identical syringes by a pharmacist not involved in patient care or outcome assessment. Both participants and clinical staff (anesthesiologists, nurses, outcome assessors) will be blinded to treatment allocation. Emergency unblinding is allowed only in the event of severe adverse events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Remimazolam with Traumatic Orthopedic Surgery (Active Comparator): Participants in this arm receive intravenous Remimazolam sedation during regional anesthesia for traumatic orthopedic surgery. Sedation dosing follows the protocol of 5 mg IV over 1 minute with supplemental doses as needed. Propofol infusion may be used as an adjunct.
  Interventions: Drug: REMIMAZOLAM BESYLATE 2.5 Mg in 1 mL INTRAVENOUS INJECTION, POWDER, LYOPHILIZED, for SOLUTION [BYFAVO]
- Remimazolam with Non-Traumatic Orthopedic Surgery (Active Comparator): Participants receive intravenous Remimazolam sedation during regional anesthesia for elective (non-traumatic) orthopedic surgery. Sedation dosing and adjunct propofol use are consistent with the protocol.
  Interventions: Drug: REMIMAZOLAM BESYLATE 2.5 Mg in 1 mL INTRAVENOUS INJECTION, POWDER, LYOPHILIZED, for SOLUTION [BYFAVO]
- Midazolam with Traumatic Orthopedic Surgery (Active Comparator): Participants receive intravenous Midazolam sedation during regional anesthesia for traumatic orthopedic surgery. Dosing is 0.025-0.05 mg/kg IV with supplemental doses if needed. Propofol may be used as adjunct sedation.
  Interventions: Drug: Midazolam
- Midazolam with Non-Traumatic Orthopedic Surgery (Active Comparator): Participants receive intravenous Midazolam sedation during regional anesthesia for elective (non-traumatic) orthopedic surgery. Sedation dosing and propofol adjunct use follow the study protocol.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — Midazolam:
  A commonly used benzodiazepine for sedation, administered intravenously at 0.025-0.05 mg/kg with supplemental doses as required. Known for effective anxiolysis and sedation but with a longer recovery profile compared to remimazolam.
  Other Names: Dormicum, Versed, Midazolam Hydrochloride
  Arms: Midazolam with Non-Traumatic Orthopedic Surgery; Midazolam with Traumatic Orthopedic Surgery
Drug: REMIMAZOLAM BESYLATE 2.5 Mg in 1 mL INTRAVENOUS INJECTION, POWDER, LYOPHILIZED, for SOLUTION [BYFAVO] — Remimazolam:
  A novel, ultra-short-acting benzodiazepine used for procedural sedation. Administered intravenously at 5 mg over 1 minute with supplemental dosing as needed. Characterized by rapid onset and quick recovery, with minimal residual sedation.
  Other Names: ByfaByfavo, Remimazolam Besylate, Remimazolam
  Arms: Remimazolam with Non-Traumatic Orthopedic Surgery; Remimazolam with Traumatic Orthopedic Surgery

SUMMARY:
This study aims to compare two medications, Remimazolam and Midazolam, used for sedation during orthopedic surgeries performed under regional anesthesia. We want to find out which medication provides better sedation during the procedure and which one affects early recovery of brain function after surgery.

Older adults (65 years and above) undergoing surgery for bone injuries or conditions will participate. We will monitor their sedation levels, blood pressure, heart rate, side effects, and how quickly they recover after surgery. We also want to see if either medication causes fewer problems with thinking and memory shortly after surgery.

The study is designed so neither the patients nor the medical staff know which medication is being given, to ensure unbiased results. Participants will be randomly assigned to receive either Remimazolam or Midazolam.

The information gathered will help doctors choose the safest and most effective sedative for older patients undergoing orthopedic surgeries, potentially improving patient comfort and recovery.

DETAILED DESCRIPTION:
1. Background and Rationale

   * Importance of effective sedation during orthopedic surgery under regional anesthesia
   * Limitations of current sedative agents (Midazolam)
   * Potential advantages of Remimazolam (rapid onset/offset, safety profile)
   * Gaps in knowledge about cognitive outcomes post-procedure in elderly patients
2. Study Objectives

   * Primary: Compare Remimazolam vs. Midazolam effects on sedation and early cognitive recovery
   * Secondary: Hemodynamics, recovery time, adverse events, patient satisfaction
3. Study Design

   * Prospective, randomized, double-blind, 2x2 factorial
   * Four arms: Remimazolam/traumatic, Remimazolam/non-traumatic, Midazolam/traumatic, Midazolam/non-traumatic
   * Single-center study
4. Patient Population and Inclusion/Exclusion Criteria

   * Age, surgery type, cognitive baseline, health status
5. Intervention Details

   * Drug dosing protocols
   * Use of adjunct propofol
   * Blinding and randomization procedures
6. Outcome Measures

   * Primary and secondary endpoints
   * Timing and methods of cognitive assessment (CAM-ICU)
   * Hemodynamic monitoring
   * Recording adverse events
7. Data Collection and Monitoring

   * Schedule of assessments
   * Safety monitoring by DSMB
   * Data confidentiality and storage
8. Statistical Analysis Plan

   * Sample size rationale
   * Statistical methods for primary and secondary outcomes
   * Handling of missing data and confounders
9. Significance and Impact

   * Potential to improve sedation choice in elderly orthopedic patients
   * Benefits for patient safety, recovery quality, and healthcare resources

Sample Detailed Description Text (expand with specifics and references):

Background and Rationale

Orthopedic surgeries in elderly patients often require sedation alongside regional anesthesia to ensure patient comfort and procedural success. Midazolam, a commonly used benzodiazepine, has a well-known sedative profile but is associated with prolonged sedation and cognitive impairment postoperatively in some cases. Remimazolam is a newer ultra-short-acting benzodiazepine with rapid onset and offset, potentially offering better control over sedation depth and faster cognitive recovery.

Currently, limited data exist comparing these agents in the context of orthopedic surgery, especially among older adults who are at higher risk for postoperative cognitive dysfunction. This study aims to fill this gap by rigorously comparing remimazolam and midazolam in a controlled clinical trial setting.

Objectives

The primary objective is to evaluate the impact of remimazolam versus midazolam on periprocedural sedation quality and early postoperative cognitive function, measured by the Confusion Assessment Method (CAM) within 72 hours after surgery.

Secondary objectives include assessment of hemodynamic stability, recovery profiles, incidence of adverse events, difficulty in spinal puncture, and patient satisfaction.

Study Design

This is a prospective, randomized, double-blind, 2x2 factorial trial conducted at the Clinical Emergency Hospital of Bucharest. Patients aged 65 and older undergoing traumatic or non-traumatic orthopedic surgery under regional anesthesia will be randomized into one of four groups.

Interventions

Patients will receive either remimazolam or midazolam following standardized dosing protocols. Propofol will be administered as an adjunct for maintenance sedation, with doses recorded and analyzed.

Outcome Measures

Primary outcomes include CAM scores assessed at multiple postoperative time points. Secondary outcomes include detailed monitoring of blood pressure, heart rate, time to full orientation, PACU stay length, adverse event rates, and subjective patient satisfaction via Likert scales.

Data Collection and Monitoring

Safety and efficacy data will be collected by blinded assessors. An independent Data and Safety Monitoring Board will oversee study progress and patient safety.

Statistical Analysis

Sample size calculations anticipate enrolling 120 participants, ensuring adequate power to detect clinically relevant differences in cognitive outcomes. Data will be analyzed using ANOVA, Kaplan-Meier, and regression models as appropriate.

Significance

This trial aims to provide evidence to guide sedative choice in elderly orthopedic patients, balancing effective sedation with cognitive safety, potentially improving patient outcomes and healthcare delivery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older.
* Scheduled for traumatic or non-traumatic orthopedic surgery under regional anesthesia.
* Able to provide informed consent or have a legally authorized representative provide consent.

Exclusion Criteria:

* Patient refusal to participate.
* Mini-Cog score less than 3 (indicative of significant cognitive impairment).
* Severe hepatic or renal failure.
* Known allergy to benzodiazepines or propofol.
* History of benzodiazepine dependence.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Early postoperative cognitive function assessed by the Confusion Assessment Method (CAM) score | 24 to 72 hours after surgery
  Cognitive function will be evaluated using the Confusion Assessment Method (CAM) to detect delirium and acute cognitive changes between 24 and 72 hours postoperatively. This tool assesses acute confusion and cognitive impairment to determine the impact of remimazolam vs. midazolam sedation on early postoperative cognition.
  Unit of Measure: CAM score (binary outcome: presence or absence of delirium) Scale Information: CAM is a diagnostic algorithm (Yes/No criteria). A positive CAM indicates the presence of delirium.

SECONDARY OUTCOMES:
Intraoperative blood pressure | Intraoperative period up to 72 hours post-surgery
  Systolic and diastolic blood pressure will be monitored intraoperatively to assess hemodynamic stability during sedation.
  Unit of Measure: mmHg
Intraoperative heart rate | Intraoperative period and up to 72 h postoperative
  Heart rate will be monitored to assess the effect of sedation on cardiovascular parameters.
  Unit of measure: Beats per minute (bpm)
Vasopressor requirement | Intraoperative period and up to 72h postoperative
  Dose and duration of vasopressors used during surgery will be recorded. Unit of Measure: μg/kg/min
Time to full orientation after surgery | Post-anesthesia care unit (PACU) period
  Time taken for the patient to become fully oriented postoperatively will be measured. Unit of Measure: Minutes
Length of stay in PACU | Post-anesthesia care unit (PACU) period
  Total duration of PACU stay postoperatively will be recorded. Unit of Measure: Minutes
Spinal Puncture Difficulty Score | During spinal puncture
  Degree of difficulty encountered during spinal anesthesia, based on a 0-5 scale. Unit of Measure: Score (0-5; higher = more difficult)
Postoperative pain (VAS score) | 0-72 hours postoperatively
  Pain will be measured using the Visual Analog Scale at multiple time points up to 72 hours. VAS score (0-10; higher = worse pain)
Patient satisfaction | Up to 72 hours postoperatively
  Patient satisfaction with anesthesia and perioperative care will be rated using a 5-point Likert scale. Unit of Measure: Likert score (1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Mirea, Associate Professor, MD, Principal Investigator — Clinical Emergency Hospital of Bucharest; Ana Maria Dumitriu, MD, PhD, Study Director — Clinical Emergency Hospital of Bucharest
Locations (1):
- Clinical Emergency Hospital of Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No
At this time, individual participant data (IPD) will not be shared due to concerns about patient privacy, data confidentiality, and institutional policies. Data sharing may be reconsidered in the future based on study results and evolving regulations.